CLINICAL TRIAL: NCT05461235
Title: A Prospective, Open, Single-arm Phase II Clinical Study to Evaluate the Efficacy and Safety of Anti-PD-1 Antibody Combined With Autologous DC and NK Cells in the Treatment of Digestive Carcinoma.
Brief Title: Anti-PD-1 Antibody Combined With Autologous DC and NK Cells in the Treatment of Digestive Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: China Medical University, China (Other)
Responsible Party: Principal Investigator, Yunpeng Liu, Director of Department of Medical Oncology, China Medical University, China
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: COMBINE
Record Dates: First submitted 2022-07-14; First posted 2022-07-18 (Actual); Last update posted 2022-07-18 (Actual); Status verified 2022-07

CONDITIONS: PD-1 Antibody; DC-Cell; NK-Cell; Gastrointestinal Tumours
MeSH Terms: interventions — pembrolizumab; Nivolumab; sintilimab; toripalimab; camrelizumab; tislelizumab

STUDY DESIGN:
Intervention Model Description: Single Group Assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Anti-PD-1 antibody combined with autologous DC and NK cells (Experimental): Anti-PD-1 antibodies (one of six options)
  1. Pembrolizumab: 2 mg/kg or 200 mg by intravenous infusion every 3 weeks
  2. Nivolumab:3 mg/kg or 240 mg by intravenous infusion every 2 weeks
  3. Sintilimab: 200 mg by intravenous infusion every 3 weeks
  4. Toripalimab: 3 mg/kg or 240 mg by intravenous infusion every 2 weeks
  5. Camrelizumab: 200 mg by intravenous infusion every 2 or 3 weeks, or 3 mg/kg by intravenous infusion every 3 weeks
  6. Tislelilzumab: 200mg by intravenous infusion every 3 weeks. DC, NK cells. 50ml of peripheral blood is collected 1 day before the dosing cycle for in vitro isolation and expansion of DC and NK cells; the first infusion of DC and NK cells (not less than 1x10^6 cells/Kg) is completed on day 14.
  Interventions: Drug: Pembrolizumab; Drug: Nivolumab; Drug: Sintilimab; Drug: Toripalimab; Drug: Camrelizumab; Drug: Tislelizumab; Biological: NK-Cell or DC-Cell

INTERVENTIONS:
Drug: Pembrolizumab — 2mg/kg or 200mg,iv,q3w
  Other Names: Keytruda
Drug: Nivolumab — 3mg/kg or 240mg,iv,q2w
  Other Names: Opdivo
Drug: Sintilimab — 200mg,iv,q3w
  Other Names: Daboshu
Drug: Toripalimab — 3mg/kg or 240mg,iv,q2w
  Other Names: Tuoyi
Drug: Camrelizumab — 200mg,iv,q2w or q3w;3mg/kg,iv,q3w
  Other Names: Airuika
Drug: Tislelizumab — 200mg,iv,q3w
  Other Names: Baizean
Biological: NK-Cell or DC-Cell — 50ml of peripheral blood was collected 1 day before the dosing cycle for in vitro isolation and amplification of DC and NK cells; the first transfusion of DC and NK cells (not less than 1x10^6 cells/Kg) was completed on day 14.

SUMMARY:
This is a prospective, open, single-arm Phase II clinical study to evaluate the efficacy and safety of anti-PD-1 antibody combined with autologous DC and NK cells in the treatment of digestive carcinoma.

DETAILED DESCRIPTION:
This is a prospective, open, single-arm Phase II clinical study to evaluate the efficacy and safety of anti-PD-1 antibody combined with autologous DC and NK cells in the treatment of digestive carcinoma.

This project aims to enhance the anti-tumour activity of DC/NK cells in combination with anti-PD-1 antibodies, and ultimately activate the patient's own immune function to improve the quality of life and survival time of tumour patients, and provide objective evidence for the widespread use of targeted immune cell therapy in the clinical setting.

ELIGIBILITY:
Inclusion Criteria:

-1. age: 18-70 years, of either sex 2. pathologically confirmed locally advanced or metastatic gastrointestinal tumour (stage III or IV according to AJCC 8th edition staging) with at least one measurable lesion (meeting RECIST 1.1 criteria) 3. ECOG PS: 0-1 points 4. have adequate organ and bone marrow function, i.e. meet the following criteria.

1. Routine blood test criteria to be met.

   1. HB ≥ 90g/L.
   2. ANC ≥1.5×109/L.
   3. PLT ≥90 x 109/L.
   4. Absolute value of lymphocytes + monocytes >2.0*10^9/L.
2. Biochemical tests are required to meet the following criteria.

   1. Total bilirubin ≤ 1.5 times the upper limit of normal (ULN).
   2. ALT and AST ≤ 2.5ULN.
   3. serum Cr ≤ 1 ULN and endogenous creatinine clearance > 60 ml/min (Cockcroft-Gault formula).

      5. international normalised ratio (INR) ≤ 1.5 and partial thromboplastin time (PPT or APTT) ≤ 1.5 ULN within 7 days prior to enrolment 6. expected survival of ≥ 3 months. 7. signed informed consent form (ICF) prior to study enrolment. 8 Women of childbearing potential must have had a pregnancy test (serum or urine) within 7 days prior to enrolment and have a negative result. Female patients of childbearing age or male patients whose sexual partners are women of childbearing age are required to use effective contraception throughout the treatment period and for 6 months after the last dose.

      Exclusion Criteria:
      * 1. known hypersensitivity to any of the components of the anti-PD-1 antibody formulation; or previous severe allergic reactions to other monoclonal antibodies.

        2. diagnosis of other malignancies, excluding radically treated basal cell carcinoma of the skin, squamous cell carcinoma of the skin and/or radically resected carcinoma in situ, within 5 years prior to the first dose 3. Subjects who have been treated with an antitumour vaccine or other antitumour agents with immunostimulatory effects (interferon, interleukin, thymidine, immune cell therapy, etc.) within 1 month prior to the first dose.

        4. CNS metastases with symptoms. Subjects may be enrolled in the study if their CNS metastases have been treated, e.g., clinical stability (MRI detection) has been maintained for at least 4 weeks, and the subject's clinical symptoms, such as neurological symptoms, are able to return to baseline levels at least 2 weeks prior to the first dose (except for residual signs or symptoms related to CNS treatment). In addition, subjects receiving stable or tapered doses of ≤10 mg/day of prednisone (or equivalent) for at least 2 weeks for clinical symptoms associated with treatment with corticosteroids are not eligible for enrollment in the study, otherwise they cannot be enrolled.

        5. Acute or chronic active hepatitis B (defined as positive HBsAg for hepatitis B virus surface antigen at screening) or hepatitis C infection. Patients with previous hepatitis B virus (HBV) infection or cured HBV infection (defined as hepatitis B core (HBc) antibody positive and HBsAg negative) who are negative for HBV DNA only may be enrolled in this study. HBV DNA testing must be performed on this group of patients prior to enrolment. Patients who are positive for hepatitis C virus (HCV) antibodies and negative for HCV RNA only by polymerase chain reaction may be enrolled in the study. Patients who are antigen-positive but have DNA/RNA copy numbers within the permissible range should be considered for antiviral treatment if enrolled in this study and DNA/RNA levels should be monitored in real time for the duration of the study.

        6. previous and current history of pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, drug-related pneumonia, severely impaired lung function and other lung diseases.

        7. active tuberculosis (TB), on anti-TB treatment or who have received anti-TB treatment within 1 year prior to the first dose 8. Human immunodeficiency virus (HIV) infected (HIV-positive), known syphilis infection 9. Patients who are considered to be at high medical risk due to severe, uncontrollable disease, non-metastatic systemic disease or having an active, uncontrollable infection. Some examples include, but not all, uncontrolled ventricular arrhythmias, recent (within 3 months) myocardial infarction, uncontrollable grand mal seizures, unstable spinal cord compression, superior vena cava syndrome, HRCT suggestive of extensive bilateral interstitial lung disease or any mental illness that may prevent informed consent from being obtained 10. active autoimmune disease requiring systemic therapy (e.g. use of disease-relieving drugs, corticosteroids or immunosuppressants) that occurred within 2 years prior to the first dose Alternative therapies (e.g. thyroxine, insulin or physiological corticosteroids for adrenal or pituitary insufficiency, etc.) are permitted Known history of primary immunodeficiency. Patients with positive autoimmune antibodies only need to confirm the presence of autoimmune disease at the discretion of the investigator.

        11. Use of immunosuppressive drugs within 4 weeks prior to first dose, excluding topical glucocorticoids by nasal spray, inhalation or other routes or physiological doses of systemic glucocorticoids (i.e. not more than 10 mg/day prednisone or equivalent doses of other glucocorticoids), temporary use of glucocorticoids for the treatment of symptoms of dyspnea in conditions such as asthma, chronic obstructive pulmonary disease is permitted.

        12. exclude subjects who have undergone major surgical procedures within 4 weeks prior to first dose, non-thoracic radiation therapy >30 Gy within 4 weeks prior to first dose, chest radiation >30 Gy within 24 weeks prior to first dose, and palliative radiation <30 Gy within 2 weeks prior to first dose who have not recovered from the toxicity and/or complications of these interventions to NCI-CTC AE ≤1 degree (except alopecia and fatigue excluded) in subjects. Palliative radiotherapy for symptom control is permitted and must be completed at least 2 weeks prior to the start of treatment with the study drug and no additional radiotherapy is planned for the same lesion. For patients who have received radiotherapy prior to 2 weeks prior to the first dose, all of the following conditions must be met for enrolment: absence of any current radiotherapy-related toxic effects, no need for glucocorticoids, exclusion of radiation pneumonia, radiation hepatitis, radiation enteritis, etc.

        13. Pregnant or breastfeeding women. 14. Participated in a clinical trial of another drug within four weeks. 15. Not considered suitable for inclusion by the investigator. Exclude subjects with a history or current evidence of any disease, treatment or laboratory abnormality that may confound the results of the study, interfere with the subject's participation in the study procedures or is not in the best interest of the subject's participation in the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Estimated)
Dates: Start 2022-07-15 (Estimated); Primary Completion 2025-07-15 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival (PFS) | one year
  PFS, defined as the time from randomization to the first occurrence of disease progression as determined by the investigator with use of RECIST v1.1 or death from any cause, whichever occurs first.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | one year
  ORR, determined using RECIST v1.1, defined as best overall response (CR or PR) across all assessment time points during the period from enrolment to termination of trial treatment.
Disease Control Rate (DCR) | one year
  Determined using RECIST v1.1 criteria.
Overall Survival (OS) | two years
  Duration from the date of initial treatment to the date of death due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Yunpeng Liu, PhD, Principal Investigator — First Hospital of China Medical University

IPD SHARING:
Plan to Share IPD: No